CLINICAL TRIAL: NCT06909643
Title: Development and Prospective Validation of a Multimodal Fusion Artificial Intelligence Model for Predicting the Efficacy of Neoadjuvant Treatment of Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-738-01
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Neoadjuvant Therapy
Keywords: Artificial Intelligence; Multimodal Fusion; Therapy Prediction; Magnetic Resonance Imaging; Digital Pathology
MeSH Terms: conditions — Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological slides of formalin-fixed, paraffin-embedded tumors resected from patients with bladder cancer undergoing radical tumor resection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bladder cancer undergoing neoadjuvant therapy: Patients pathological diagnosed with bladder cancer undergoing neoadjuvant therapy.
  Interventions: Diagnostic Test: Artificial intelligence (AI)-based diagnostic model

INTERVENTIONS:
Diagnostic Test: Artificial intelligence (AI)-based diagnostic model — Collect magnetic resonance imaging and pathological slides of resected tumor of the enrolled patients. Analyze the data using the AI model to generate diagnostic results (sensitive or insensitive to the neoadjavant therapy). No intervention to patients would be performed in this diagnostic test study.

SUMMARY:
This study is a multi-center observational study without interventions, including the construction of an AI diagnostic model and retrospective testing of a multi-center cohort. The study participants are bladder cancer patients who have undergone imaging examinations, been pathologically diagnosed, and received neoadjuvant treatment, with complete clinical and pathological data. The study plans to enroll 130 patients from our center, collecting corresponding imaging images, and gathering clinical and genomic data to build and internally validate a multimodal AI model. The model's generalization and robustness will be tested to explore the association between multimodal data and the efficacy of neoadjuvant treatment for bladder cancer. The aim is to assist clinicians in predicting and evaluating the efficacy of neoadjuvant treatment for bladder cancer, with the goal of improving patient diagnosis, treatment outcomes, and prognosis.

DETAILED DESCRIPTION:
Bladder cancer is one of the most common malignancies of the genitourinary system worldwide. For muscle - invasive bladder cancer amenable to radical resection, the standard treatment is neoadjuvant therapy combined with radical cystectomy, with neoadjuvant therapy playing a crucial role. Currently, numerous studies have shown that cisplatin - based neoadjuvant chemotherapy can downstage tumors, reduce the risk of mortality in bladder cancer patients, improve survival rates, and enhance prognosis. Other treatment approaches such as neoadjuvant immunotherapy, targeted therapy, and combination therapies are also under investigation. However, responses to neoadjuvant therapy vary among bladder cancer patients, with some not achieving the desired therapeutic goals. Therefore, accurately predicting participants' response to treatment can provide an important reference for personalized and precise treatment of bladder cancer.

In recent years, as advancements in computational power and data storage capacity, artificial intelligence (AI) has been widely applied in the field of digital diagnostics. AI technologies can extract and integrate a large number of features from multimodal data such as pathology, imaging, and clinical records, enabling precise disease diagnosis, prognosis assessment, and treatment prediction. In the field of tumor treatment prediction, multimodal AI technologies have achieved numerous breakthroughs, developing efficacy prediction models for tumors such as rectal and breast cancer based on imaging and pathological data, and validating the models' generalization capabilities through external validation.

Therefore, the investigators plan to construct and validate a "Bladder Cancer Neoadjuvant Treatment Efficacy Prediction Model" based on multimodal data such as MRI images, digital pathology images, and clinical records of bladder cancer patients, and develop an AI - assisted prediction software for neoadjuvant treatment efficacy in bladder cancer. The investigators hope that this AI diagnostic model can serve as an auxiliary tool to assist clinicians in stratifying neoadjuvant treatment efficacy in bladder cancer patients, thereby formulating precise treatment plans, reducing the consumption of human and material resources, and seizing the optimal treatment opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Bladder occupying lesions, with histopathological confirmation of bladder cancer after resection.
* Planned neoadjuvant therapy and radical cystectomy.

Exclusion Criteria:

* Patients who have not undergone standard bladder imaging examinations or have missing imaging or pathological data.
* Patients who have received local treatments (such as interventional embolization) or systemic treatments (such as radiotherapy, chemotherapy, immunotherapy, or targeted therapy).
* Poor quality of imaging or pathological images.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed bladder cancer who undergo neoadjuvant therapy and radical cystectomy are planned to be enrolled in this diagnostic test to assess the model's clinical application capability.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity | For each enrolled patient, the diagnosis results of AI model will be obtained in several days after neoadjuvant therapy, and the sensitivity of the AI model will be evaluated through study completion, an average of 3 year.
  the number of correctly diagnosed positive patient (sensitive to therapy), to be divided by the number of patients in total.

SECONDARY OUTCOMES:
specificity | For each enrolled patient, the diagnosis results of AI model will be obtained in several days after neoadjuvant therapy, and the specificity of the AI model will be evaluated through study completion, an average of 3 year.
  the number of correctly diagnosed negative patients (therapy insensitive), to be divided by the number of negative patients in total.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, magnetic resonance imaging, pathological slide images and other patient-related data are not publicly accessible.